CLINICAL TRIAL: NCT03815162
Title: Pilot Study to Investigate the Effect of Cocoa Flavanols on Symptoms in Primary Raynaud's Phenomenon
Brief Title: Cocoa Flavanol Supplementation in Raynaud's Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Elizabeth Simpson, Senior Research Fellow, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 112-1809
Record Dates: First submitted 2019-01-18; First posted 2019-01-24 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Primary Raynaud Phenomenon
Keywords: cocoa flavanols

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo controlled study. Block randomised with equal allocation of participants between groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Opaque capsules of equal size and appearance presented in similar bottles labelled only by a code. Code to product information is held by the manufacturer and un-blinding of the PI will only occur once the study analysis has been completed or in the event of a serious adverse event occurring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flavanol Cocoa extract (Experimental): 278mg total flavanols (38.3mg epicatechin) per opaque cellulose capsule 3 capsules consumed once per day (836 mg total flavanols; 115mg epicatechin) for 3 months
  Interventions: Dietary Supplement: High Flavanol Cocoa extract
- Alkalised cocoa (Placebo Comparator): 0mg total flavanols (0mg epicatechin) per opaque cellulose capsule 3 capsules consumed once per day (0mg total flavanols; 0mg epicatechin) for 3 months
  Interventions: Dietary Supplement: Alkalised cocoa

INTERVENTIONS:
Dietary Supplement: High Flavanol Cocoa extract — Experimental group
  Arms: High Flavanol Cocoa extract
Dietary Supplement: Alkalised cocoa — Control group
  Arms: Alkalised cocoa

SUMMARY:
The study aims to investigate the effect that supplementing the diet with cocoa flavanols has on vasospasm symptoms and temperature regulation in women with primary Raynaud's phenomenon (PRP). Participants will be randomised to consume either high flavanol cocoa extract or low flavanol cocoa (placebo) daily for 3 months.

DETAILED DESCRIPTION:
Primary Raynaud's phenomenon (PRP) is characterised by periodic vasospasm of the fingers and toes precipitated by exposure to cold or emotional stimuli and stress. Previous studies have demonstrated that underlying this condition there can be vascular endothelium dysfunction. Pharmacological interventions used to relieve symptoms and complications in PRP include drugs targeted at increasing nitric oxide (NO; transdermal nitrates) levels. Cocoa derived products, rich in the phytonutrients 'flavanols', have been shown to increase the bioavailability of NO at the vascular endothelium and promote vasodilation, which may address an underlying cause of PRP and mitigate symptoms. Previous work carried out in the research group has indicated that the acute consumption of cocoa does not compromise the counter-regulatory responses to localised cold exposure in those with PRP.

30 individuals with PRP will be recruited. Those interested in taking part will attend a medical screening and consent visit. If recruited, a participant number will be assigned to them sequentially and they will be randomised to either experimental or control group, with neither the participants nor the research team knowing which group they have been allocated to. Participants will be asked to complete a diet diary before attending 4 further visits over a period of 3 months.

Visit 1 (pre-intervention) and 4 (end of intervention); immediately on arrival, participants will be asked to lie semi-supine on a hospital bed. Skin temperature (surface thermocouples) and 'core' temperature (infrared tympanic thermometer) will start to be recorded to identify when these parameters have stabilized in room temperature (set at 25oC). Blood pressure will be taken using an arm cuff. Then a Finometer cuff will be attached to the left middle finger to record cardiovascular parameters (Blood pressure /heart rate/ cardiac output) and a laser Doppler probe will be attached to the dorsum of both index fingers to assess skin blood flow. Once the finger skin temperature has remained stable for 6 minutes, baseline Finometer and laser Doppler measurements will be recorded and the skin and 'core' temperature will be noted. Then, the right hand will be placed in a temperature regulated box which is set at an air temperature of 0oC. The hand will be cooled to a finger skin temperature of 15oC, then the box temperature will be modified to maintain the skin temperature at 15oC. The time that it takes for the skin temperature on the fingers to reach 15oC will be recorded. With the finger skin temperature stable at 15oC, Finometer and laser Doppler measurements will be repeated and the 'core' temperature at this point noted. Then, the hand will be removed from the chamber, and allowed to equilibrate in room temperature. The time taken for the skin temperature to reach stability will be recorded, as will the absolute temperature that it stabilises to. Measures above will be repeated once hand temperature is stable. Once these measures have been made, all equipment will be removed and a 15ml blood sample will be taken (for epicatechin, glucose and insulin analysis). The participant will be asked to complete 3 questionnaires (SF-36, Raynaud's symptoms and a food frequency questionnaire). Participants will also return a 4-day diet diary at visits 1 and 4, and their symptom diary at visit 4.

Visits 2 (end of month 1) and 3 (end of month 2); participants will return a 4-day diet diary, symptom diary and any unused capsules. They will also have a resting blood pressure measurement made, weight measured and be asked to complete 3 questionnaires (SF-36, Raynaud's symptoms and a food frequency questionnaire).

At the end of Visits 1, 2 and 3, participants will be given a months' supply of capsules, a symptom diary and a diet diary (to be completed in the week prior to the next visit).

ELIGIBILITY:
Inclusion Criteria:

* Experience symptoms of Primary Raynaud's Phenomenon, with >1 attack / week through the winter months
* Daily consumption of caffeine containing foods/drinks.
* BMI <27kg/m2

Exclusion Criteria:

* pregnant or breast feeding (women only),
* clinically significant metabolic or endocrine abnormalities
* fasting glucose >6.5mmol/l,
* taking Bosentan, aspirin, dipyridamole, heparin or transdermal nitrates,
* herbal supplement use,
* food allergies related to the investigational product (cocoa, peanuts, milk),
* sensitivity to methylxanthines (e.g. caffeine, theobromine).
* Presence or history of digital ulceration,
* blood parameters suggesting secondary Raynaud's,
* history of migraines

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Vasospasm | 3 months
  frequency of vasospasm

SECONDARY OUTCOMES:
Severity of vasospasm symptoms | 3 months
  visual analogue score for pain associated with each vasospasm occasion. Participants indicate pain intensity by placing a vertical line on a 100mm horizontal line where the start of the line (left-hand side; 0mm) represents 'no pain' and the end of the line (right-hand side; 100mm) represents 'most severe pain'. Distance of the vertical line from 0 provides the visual analogue score. A lower score indicates a more favourable outcome.
Duration of vasospasm symptoms | 3 months
  duration that symptoms persist for on each vasospasm occasion
Raynaud's Condition score | 3 months
  Assessment of Raynaud's symptoms using the validated Raynaud's Condition Score. This is a 1 to 10 Likert scale, with 0 representing 'no difficulty' and 10 indicating 'extreme difficulty' with symptoms; collected daily for 3 months, a lower score indicates a more favourable outcome.
Blood pressure | pre-intervention
  blood pressure measured by automated oscillometric blood pressure
Blood pressure | 4 weeks after starting intervention
  blood pressure measured by automated oscillometric blood pressure
Blood pressure | 8 weeks after starting intervention
  blood pressure measured by automated oscillometric blood pressure
Blood pressure | 12 weeks after starting the intervention
  blood pressure measured by automated oscillometric blood pressure
Dietary polyphenol intake | pre-intervention
  estimation of dietary polyphenols made by food frequency questionnaire
Dietary polyphenol intake | 4 weeks after starting intervention
  estimation of dietary polyphenols made by food frequency questionnaire
Dietary polyphenol intake | 8 weeks after starting intervention
  estimation of dietary polyphenols made by food frequency questionnaire
Dietary polyphenol intake | 12 weeks after starting the intervention
  estimation of dietary polyphenols made by food frequency questionnaire
Ambient skin temperature | pre-intervention
  skin temperature of a finger exposed to an environmental temperature of 25oC, before cooling
Ambient skin temperature | 12 weeks after starting the intervention
  skin temperature of a finger exposed to an environmental temperature of 25oC, before cooling
Ambient skin blood flow | pre-intervention
  finger blood flow (measured using laser Doppler flowmetry) when exposed to an environmental temperature of 25oC, before cooling
Ambient skin blood flow | 12 weeks after starting the intervention
  finger blood flow (measured using laser Doppler flowmetry) when exposed to an environmental temperature of 25oC, before cooling
Skin temperature response to acute cooling | pre-intervention
  The time taken for skin temperature of the finger to stabilise in response to localised cooling (in an air temperature of 0oC)
Skin temperature response to acute cooling | 12 weeks after starting the intervention
  The time taken for skin temperature of the finger to stabilise in response to localised cooling (in an air temperature of 0oC)
Skin blood flow response to acute cooling | pre-intervention
  Finger Skin blood flow; measurement (using laser Doppler flowmetry) made once finger skin temperature has stabilised in response to localised cooling (in an air temperature of 0oC)
Skin blood flow response to acute cooling | 12 weeks after starting the intervention
  Finger Skin blood flow; measurement (using laser Doppler flowmetry) made once finger skin temperature has stabilised in response to localised cooling (in an air temperature of 0oC)
Skin temperature response to re-warming | pre-intervention
  The time taken for skin temperature of finger to stabilise in an environmental temperature of 25oC following localised cooling (in an air temperature of 0oC)
Skin temperature response to re-warming | 12 weeks after starting the intervention
  The time taken for skin temperature of finger to stabilise in an environmental temperature of 25oC following localised cooling (in an air temperature of 0oC)
Skin temperature after re-warming | pre-intervention
  skin temperature that a finger exposed to an environmental temperature of 25oC stabilises to after localised cooling
Skin temperature after re-warming | 12 weeks after starting the intervention
  skin temperature that a finger exposed to an environmental temperature of 25oC stabilises to after localised cooling
Quality of life score | pre-intervention
  Assessed using SF-36 questionnaire. Responses are coded and normalised to the UK population, as per standard methods, and a score for mental and physical health calculated; a higher score indicating a more favourable outcome
Quality of life score | 4 weeks after starting intervention
  Assessed using SF-36 questionnaire. Responses are coded and normalised to the UK population, as per standard methods, and a score for mental and physical health calculated; a higher score indicating a more favourable outcome
Quality of life score | 8 weeks after starting intervention
  Assessed using SF-36 questionnaire. Responses are coded and normalised to the UK population, as per standard methods, and a score for mental and physical health calculated; a higher score indicating a more favourable outcome
Quality of life score | 12 weeks after starting the intervention
  Assessed using SF-36 questionnaire. Responses are coded and normalised to the UK population, as per standard methods, and a score for mental and physical health calculated; a higher score indicating a more favourable outcome
Attrition rate | 2 years
  Number of participants completing the protocol as a proportion of those who were randomised to the study
Adverse events | 3 months
  Any injury, accident or illness experienced over the intervention period will be documented
Recruitment rate | 2 years
  number of people volunteering to take part in the study as a proportion of those expressing initial interest

CONTACTS AND LOCATIONS:
Overall Officials: Ian A Macdonald, PhD, Study Director — University of Nottingham
Locations (1):
- David Greenfield Human Physiology Laboratories, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared with other researchers

REFERENCES:
- [Background] Herrick A. Raynaud's phenomenon. Curr Treat Options Cardiovasc Med. 2008 Apr;10(2):146-55. doi: 10.1007/s11936-008-0016-y. PMID 18325317
- [Background] Chung L, Shapiro L, Fiorentino D, Baron M, Shanahan J, Sule S, Hsu V, Rothfield N, Steen V, Martin RW, Smith E, Mayes M, Simms R, Pope J, Kahaleh B, Csuka ME, Gruber B, Collier D, Sweiss N, Gilbert A, Dechow FJ, Gregory J, Wigley FM. MQX-503, a novel formulation of nitroglycerin, improves the severity of Raynaud's phenomenon: a randomized, controlled trial. Arthritis Rheum. 2009 Mar;60(3):870-7. doi: 10.1002/art.24351. PMID 19248104